CLINICAL TRIAL: NCT02309424
Title: The Effect of Vinegar on Glucose and Lipid Metabolism in Peripheral Tissues in Subjects With Impaired Glucose Tolerance or Type 2 Diabetes
Brief Title: The Effect of Vinegar on Glucose and Lipid Metabolism in Subjects With Impaired Glucose Tolerance or Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Collaborators: Hellenic National Diabetes Center (Other)
Responsible Party: Principal Investigator, Panayota Mitrou, Senior Researcher, MD, PhD, Attikon Hospital
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 167/11-06-08
Record Dates: First submitted 2014-12-01; First posted 2014-12-05 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vinegar (Active Comparator): 0,50mmol vinegar (6% acetic acid)
  Interventions: Dietary Supplement: Vinegar
- Placebo (Placebo Comparator): 50 ml water
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vinegar — 0,50mmol vinegar (6% acetic acid)
  Arms: Vinegar
Other: Placebo — 50 ml water
  Arms: Placebo

SUMMARY:
This open, randomized, cross-over, placebo-controlled study aims to investigate the effects of vinegar on glucose metabolism, endothelial function and circulating lipid levels in subjects with impaired glucose tolerance or type 2 diabetes, using the arteriovenous difference technique.

DETAILED DESCRIPTION:
Subjects with IGT or type 2 diabetes will be randomised to consume 20ml vinegar (6% acetic acid) or placebo before a mixed meal. Plasma samples will be taken for 300min from the radial artery and from a forearm vein for measurements of glucose, insulin, triglycerides, non-esterified fatty acids (NEFA) and glycerol. Muscle blood flow will be measured with strain-gauge plethysmography. Glucose flux will be calculated as the arteriovenous difference of glucose multiplied by the blood flow rates.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with impaired glucose tolerance or newly diagnosed type 2 diabetes before the initiation of medication therapy
2. Recreationally active
3. With stable body weight and diet during the last two months.

Exclusion Criteria:

1. Any systemic disease (besides glucose abnormalities)
2. Any medication therapy
3. Diabetic complications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-07; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Muscle glucose uptake following meal ingestion (area under the glucose uptake versus time curve-AUC) | 0, 30, 60, 90, 120, 180, 240, 300 min postmeal

SECONDARY OUTCOMES:
Plasma glucose levels following meal ingestion (area under the plasma concentration versus time curve-AUC) | 0, 30, 60, 90, 120, 180, 240, 300 min postmeal
Plasma insulin levels following meal ingestion (area under the plasma concentration versus time curve-AUC) | 0, 30, 60, 90, 120, 180, 240, 300 min postmeal
Plasma triglyceride levels following meal ingestion (area under the plasma concentration versus time curve-AUC) | 0, 30, 60, 90, 120, 180, 240, 300 min postmeal
Plasma NEFA levels following meal ingestion (area under the plasma concentration versus time curve-AUC) | 0, 30, 60, 90, 120, 180, 240, 300 min postmeal
Plasma glycerol levels following meal ingestion (area under the plasma concentration versus time curve-AUC) | 0, 30, 60, 90, 120, 180, 240, 300 min postmeal
Muscle blood flow following meal ingestion (area under the blood flow rates versus time curve-AUC) | 0, 30, 60, 90, 120, 180, 240, 300 min postmeal
Number of participants with adverse events | 300 min postmeal

CONTACTS AND LOCATIONS:
Overall Officials: George D Dimitriadis, Professor, Study Director — Attikon Hospital

REFERENCES:
- [Derived] Mitrou P, Petsiou E, Papakonstantinou E, Maratou E, Lambadiari V, Dimitriadis P, Spanoudi F, Raptis SA, Dimitriadis G. Vinegar Consumption Increases Insulin-Stimulated Glucose Uptake by the Forearm Muscle in Humans with Type 2 Diabetes. J Diabetes Res. 2015;2015:175204. doi: 10.1155/2015/175204. Epub 2015 May 6. PMID 26064976